CLINICAL TRIAL: NCT05655702
Title: DRug Use & Infections in ViEtnam: TuBerculosis Control Towards Tuberculosis Elimination Among People Who Inject Drugs: Evaluation of a Community-based Intervention in Vietnam
Brief Title: DRug Use & Infections in ViEtnam: TuBerculosis Control
Acronym: DRIVE-TB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Haiphong University of Medicine and Pharmacy (Other); Expertise France (Other); Université Montpellier (Other); New York University (Other); CENTER FOR SUPPORTING COMMUNITY DEVELOPMENT INITIATIVES (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ANRS 0092s DRIVE-TB
Record Dates: First submitted 2022-11-02; First posted 2022-12-19 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Tuberculosis
Keywords: people who inject drug; screening
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- community-based TB intervention (Other)
  Interventions: Other: Community based TB intervention

INTERVENTIONS:
Other: Community based TB intervention — * 3 bi-annual RDSS (RDSS1, 2 and 3), for TB screening
  * A PWID-specific Information and communication (I&C) TB module to improve PWID awareness about TB,
  * Peer group support to facilitate TB treatment initiation and retention,
  * Implementation of a peer support contact tracing and screening for active TB in contacts.

SUMMARY:
The overarching purpose of the proposed research is to demonstrate that a targeted, multi-component community-based intervention among PWID in Hai Phong will decrease TB prevalence among this very high-risk population.

DETAILED DESCRIPTION:
Vietnam has a strong National TB Program (NTP), but it belongs to the 20 countries with the highest TB burden in the world. A TB prevalence study among people who inject drugs (PWID) was conducted as part of the Drug use & Infections in ViEtnam (DRIVE) program, in collaboration with a local screening initiative (Zero TB Vietnam, national TB program - NTP) in 2018 in Hai Phong. While the annual TB rate in the general population of Vietnam is 0.13%, this study found an alarming prevalence of confirmed TB cases from 1.8% to 5.6% among PWID. Some populations, such as people who inject drugs (PWID), combine a very high risk of TB and low access to TB care. Based on the investigators experience in operational research among PWID and their expertise in TB, they designed an intervention to end TB among a highly vulnerable population such as PWID, through significant community involvement.

They hypothesize that a targeted, multi-component community-based intervention among PWID in Hai Phong will decrease TB prevalence among this very high-risk population.

The DRIVE-TB intervention will use four repeated large-scale randomized driven sampling surveys (RDSS) to identify TB-infected PWID in the community. During RDSS 1 and 4 all participants will undergo a questionnaire on TB symptoms, and have CRP, chest X-ray, and sputum collection for Xpert MTB-RIF®. In RDSS 2 and 3, participants will be screened through the best screening algorithm (elaborated in RDSS1). Participants from all RDSS will also be screened for LTBI through Tuberculin Skin Test (TST). Moreover the 3HP ancillary study, a therapeutic cohort will assess the acceptability, safety, adherence, and cost of a 12-dose once-weekly regimen of isoniazid/rifapentine (3HP) to prevent TB disease among RDSS 2 participants with a positive QuantiFERON test result will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Self-declaring injecting heroin or any other drug
* Positive urine test for heroin or methamphetamine
* Presence of recent injection site marks

Exclusion Criteria:

* Unable to understand or refused to sign informed consent
* Patients currently under treatment for active TB
* Any condition which might, in the investigator's opinion, compromise the safety of the patient by participating in the study, including very severe clinical condition
* Person deprived of freedom by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence of confirmed TB cases at RDSS 1 and RDSS 4 | 2 years between RDSS 1 and 4

SECONDARY OUTCOMES:
Assess TB awareness | 2 years
  Appropriate answers to a set of questions on the knowledge of TB encompassing 3 domains (symptoms, mode of transmission, treatment), at RDSS1 and RDSS4.
The feasibility and efficacy of the TB mass screening | Through study completion, an average of 2 years
  will be evaluated by the proportion of eligible RDSS participants (i.e. meeting the inclusion criteria) who consent to participate after information. The efficacy of the mass screening, defined by the proportion of those actually tested among the RDSS participants.
Proportion of confirmed TB cases who have initiated TB treatment among those who have attended the referral TB center for confirmation in RDSS 1, 2, 3. | Up to one year
Prevalence of active TB and LTBI among PWID contacts | 1 year
The incidence of active TB and LTBI among PWID contacts at 6 and 12 months. | 2 years
The proportion of PWID contacts actually screened for TB at the community study site. | 1 year
The incidence of TB infection (LTBI and active TB) among PWID in Hai Phong | 2 years
HIV viremia prevalence at RDSS1 | At baseline
  defined by the ratio of PWID with HIV viral load >1000 copies/mL among all PWID, whatever their HIV status
Incremental cost-effectiveness ratio (ICER) and cost per DALY averted. | At baseline
Acceptability of the 3HP regimen, | 3 months after inclusion in RDSS2
  Defined by both the proportion of RDSS2 participants who accept to participate in the LTBI study after information, and by those who initiated a isoniazid/rifapentine (3HP) among those eligible (i.e. with a positive QuantiFERON test result).
Safety of the 3HP regimen, | 3 months after inclusion in RDSS2
  Defined by the rate of patients with grade ≥2 adverse events, potentially related to the 3HP regimen, including craving symptoms.
Proportion of participants who have completed a 12-dose once-weekly regimen of isoniazid/rifapentine (3HP) among those who have initiated 3HP. | 3 months after inclusion in RDSS2

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas NAGOT, Principal Investigator — PCCI UMR 1058 - INSERM, Univ Montpellier, EFS, Montpellier, Franc; Huong DUONG THI, Principal Investigator — Hai Phong University of Medicine and Pharmacy, Vietnam
Locations (2):
- Vietnam (2):
  - Hai Phong University of Medecine and Pharmacy, Haiphong
  - Viettiep 2 Hospital, Haiphong

IPD SHARING:
Plan to Share IPD: No